CLINICAL TRIAL: NCT03278769
Title: Relation Between Lung Protective Mechanical Ventilation, Intracranial Pressure, Autoregulation and Brain Oxygenation in Neurointensive Care Patients
Brief Title: Ventilator Settings on Patients With Acute Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Hôpital de la Croix-Rousse (Other)
Responsible Party: Principal Investigator, Shirin Kordasti Frisvold, Principal investigator, PhD, University Hospital of North Norway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Brain-Vent
Record Dates: First submitted 2017-08-29; First posted 2017-09-12 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Acute Brain Injury; Ventilator-Induced Lung Injury; Cerebrovascular Circulation
MeSH Terms: conditions — Brain Injuries; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ventilator setting (Experimental): Positive end-expiratory pressure , Tidal volume
  Interventions: Procedure: Lung protective ventilator settings

INTERVENTIONS:
Procedure: Lung protective ventilator settings — Positive end-expiratory pressure 12, Tidal volume 6 milliliter/kilogram predicted body weight

SUMMARY:
The present study is an explorative analysis of the relationship between cerebral blood perfusion and oxygenation and lung mechanical variables at different ventilator settings. It is a safety study excluding patients with severe lung injury or brain edema.

DETAILED DESCRIPTION:
The primary goal is to carry out baseline measurements to enable conclusions concerning the safety of lung protective ventilator settings before extending the study to patients with more severe brain and/or lung injury in the future.

The primary objective is to investigate if lung protective ventilator settings (higher Positive end-expiratory pressure and lower tidal volume) as compared with conventional settings.

1. increase intracranial pressure
2. diminish cerebral vasoreactive autoregulation as assessed by pressure reactivity index, ie pressure reactivity index will turn positive, which means that it will change the state from intact to impaired autoregulation.

The secondary objective is an exploratory analysis of the relationship between ventilator settings and other well defined respiratory, cerebral, and cardiovascular variables, including transpulmonary pressure.

ELIGIBILITY:
Inclusion Criteria:

* • Any tracheally intubated or tracheotomized adult patient with ABI with GCS< 9 on controlled ventilation requiring continuous ICP measurement.
* Proxy informed consent from relatives.

Exclusion Criteria:

* • ICP > 22 mmHg before treatment of high ICP
* Acute respiratory failure defined as partial pressure of oxygen/ inspiratory oxygen fraction (PaO2/FiO2) ratio < 40 kPa and Xray pathology
* History of pulmonary disese: Chronic respiratory failure diagnosis stage III and IV in the GOLD classification, pulmectomy, lobectomy or restrictive lung disease.
* Body mass index (BMI) > 35.
* Known right or biventricular cardiac failure with cardiac index < 2,5 L/min/m2 or ejection fracture < 40 %.
* Refractory hypovolemia as diagnosed with pulse pressure variation > 12 % with tidal volume 8 ml/predicted bodyweight (intubated on controlled ventilation) or passive leg rise test with > 10 % increase in stroke volume measured by VTI echocardiography or PICCO.
* Medulla lesion that affect the autonomic nervous system.
* Patients who has undergone decompressive craniectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Intracranial pressure | 120 minutes
  intracranial pressure increase with lung protective setting
pressure reactivity index | 120 minutes
  Diminished pressure reactivity index

CONTACTS AND LOCATIONS:
Overall Officials: Shirin K Frisvold, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smielewski P, Lavinio A, Timofeev I, Radolovich D, Perkes I, Pickard JD, Czosnyka M. ICM+, a flexible platform for investigations of cerebrospinal dynamics in clinical practice. Acta Neurochir Suppl. 2008;102:145-51. doi: 10.1007/978-3-211-85578-2_30. PMID 19388307
- [Background] Koutsoukou A, Katsiari M, Orfanos SE, Kotanidou A, Daganou M, Kyriakopoulou M, Koulouris NG, Rovina N. Respiratory mechanics in brain injury: A review. World J Crit Care Med. 2016 Feb 4;5(1):65-73. doi: 10.5492/wjccm.v5.i1.65. eCollection 2016 Feb 4. PMID 26855895
- [Background] Mauri T, Yoshida T, Bellani G, Goligher EC, Carteaux G, Rittayamai N, Mojoli F, Chiumello D, Piquilloud L, Grasso S, Jubran A, Laghi F, Magder S, Pesenti A, Loring S, Gattinoni L, Talmor D, Blanch L, Amato M, Chen L, Brochard L, Mancebo J; PLeUral pressure working Group (PLUG-Acute Respiratory Failure section of the European Society of Intensive Care Medicine). Esophageal and transpulmonary pressure in the clinical setting: meaning, usefulness and perspectives. Intensive Care Med. 2016 Sep;42(9):1360-73. doi: 10.1007/s00134-016-4400-x. Epub 2016 Jun 22. PMID 27334266
- [Derived] Beqiri E, Smielewski P, Guerin C, Czosnyka M, Robba C, Bjertnaes L, Frisvold SK. Neurological and respiratory effects of lung protective ventilation in acute brain injury patients without lung injury: brain vent, a single centre randomized interventional study. Crit Care. 2023 Mar 20;27(1):115. doi: 10.1186/s13054-023-04383-z. PMID 36941683

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03278769/Prot_SAP_000.pdf